CLINICAL TRIAL: NCT05059301
Title: A Phase 3, Randomized, Double-blind, Multi-country Study to Evaluate Consistency, Safety, and Reactogenicity of 3 Lots of RSVPreF3 OA Investigational Vaccine Administrated as a Single Dose in Adults Aged 60 Years and Above
Brief Title: A Study of 3 Lots of an Investigational Vaccine Against Respiratory Syncytial Virus (RSV) in Adults Aged 60 Years and Above
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 217131; 2021-002225-18 (EudraCT Number)
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Results first posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-01

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory syncytial virus; Adults aged 60 years and above; Lot-to-lot consistency; Safety; Reactogenicity
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study is double blind from start to final analysis after which the study is considered single blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- RSV OA_Lot 1 (Experimental): Participants received 1 dose of a combination of the RSVPreF3 antigen Lot 1 and AS01E adjuvant Lot A at Day 1 and were followed up until the study end (Month 6).
  Interventions: Biological: RSVPreF3 OA investigational vaccine
- RSV OA_Lot 2 (Experimental): Participants received 1 dose of a combination of the RSVPreF3 antigen Lot 2 and AS01E adjuvant Lot B at Day 1 and were followed up until the study end (Month 6).
  Interventions: Biological: RSVPreF3 OA investigational vaccine
- RSV OA_Lot 3 (Experimental): Participants received 1 dose of a combination of the RSVPreF3 antigen Lot 3 and AS01E adjuvant Lot C at Day 1 and were followed up until the study end (Month 6).
  Interventions: Biological: RSVPreF3 OA investigational vaccine

INTERVENTIONS:
Biological: RSVPreF3 OA investigational vaccine — One dose of a unique combination of the RSVPreF3 antigen lots (Lot 1, Lot 2 or Lot 3) and extemporaneously reconstituted with AS01E adjuvant lots (Lot A, Lot B and Lot C), administered intramuscularly in the deltoid region of the non-dominant arm, at Day 1.

SUMMARY:
The purpose of this study is to assess the lot-to-lot consistency in terms of immunogenicity and evaluate the safety and reactogenicity of 3 lots of the RSVPreF3 OA investigational vaccine administered as a single dose in adults ≥ 60 years of age (YOA).

ELIGIBILITY:
Inclusion Criteria:

* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol. A male or female ≥ 60 YOA at the time of first study intervention administration.
* Participants living in the general community or in an assisted living facility that provides minimal assistance, such that the participant is primarily responsible for self care and activities of daily living.
* Written or witnessed informed consent obtained from the participant prior to performance of any study specific procedure.
* Participants who are medically stable in the opinion of the investigator at the time of vaccination. Participants with chronic stable medical conditions with or without specific treatment, such as diabetes, hypertension or cardiac disease, can participate in this study if considered by the investigator as medically stable.

Exclusion Criteria:

Medical conditions

* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease or immunosuppressive/cytotoxic therapy, based on medical history, and physical examination (no laboratory testing required).
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention(s).
* Hypersensitivity to latex.
* Serious or unstable chronic illness.
* Any history of dementia or any medical condition that moderately or severely impairs cognition.
* Recurrent or un controlled neurological disorders or seizures. Participants with medically controlled active or chronic neurological diseases can be enrolled in the study as per investigator assessment, provided that their condition will allow them to comply with the requirements of the protocol.
* Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.

Prior/Concomitant therapy

* Use of any investigational or non registered product (drug, vaccine or medical device) other than the study intervention(s) during the period beginning 30 days before study intervention administration and ending 30 days after study intervention administration, or planned use during the study period.
* Planned or actual administration of a vaccine not foreseen by the study protocol in the period starting 30 days before and ending 30 days after the study intervention administration, with the exception of inactivated and subunit influenza vaccines which can be administered up to 14 days before or from 14 days after the study vaccination.
* Note: In case an emergency mass vaccination for an unforeseen public health threat (e.g. a pandemic) is recommended and/or organized by the public health authorities, outside the routine immunization program, the time period described above can be reduced if necessary for that vaccine provided it is used according to the local governmental recommendations and that the Sponsor is notified accordingly. Previous vaccination with an RSV vaccine.
* Administration of long acting immune modifying drugs or planned administration at any time during the study period.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 90 days before the administration of the study intervention or planned administration during the study period.
* Chronic administration (defined as more than 14 consecutive days in total) of immunosuppressants or other immune modifying drugs during the period starting 90 days prior to the study intervention administration or planned administration during the study period. For corticosteroids, this will mean prednisone ≥ 20 mg/day or equivalent. Inhaled and topical steroids are allowed.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non investigational vaccine/product (drug or invasive medical device).

Other exclusions

* History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.
* Planned move during the study period that will prohibit participating in the study until study end.
* Bedridden participants.
* Participation of any study personnel or their immediate dependents, family, or household members.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 770 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (9):
  - GSK Investigational Site, Waterbury, Connecticut
  - GSK Investigational Site, Brooksville, Florida
  - GSK Investigational Site, Immokalee, Florida
  - GSK Investigational Site, Buford, Georgia
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Petal, Mississippi
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Houston, Texas
- Canada (7):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Moncton, New Brunswick
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Sweden (3):
  - GSK Investigational Site, Eskilstuna
  - GSK Investigational Site, Karlskrona
  - GSK Investigational Site, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

REFERENCES:
- [Derived] Ferguson M, Murray A, Pliamm L, Rombo L, Sanmartin Berglund J, David MP, De Schrevel N, Maschino F, Kotb S, Olivier A, Hulstrom V. Lot-to-lot immunogenicity consistency of the respiratory syncytial virus prefusion F protein vaccine in older adults. Vaccine X. 2024 Apr 27;18:100494. doi: 10.1016/j.jvacx.2024.100494. eCollection 2024 Jun. PMID 38746060

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 770 participants enrolled 757 received the study vaccine and were included in the Exposed Set.
Period: Overall Study
Arm/Group | RSV OA_Lot 1 | RSV OA_Lot 2 | RSV OA_Lot 3
Started | 251 | 253 | 253
Completed | 249 | 248 | 248
Not Completed | 2 | 5 | 5
Not completed — Adverse Event | 0 | 2 | 2
Not completed — Lost to Follow-up | 2 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RSV OA_Lot 1 | RSV OA_Lot 2 | RSV OA_Lot 3 | Total
Number analyzed (Participants) | 251 | 253 | 253 | 757
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.7 (6.6) | 70.1 (6.6) | 69.9 (6.6) | 69.9 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 131 | 109 | 371
  Male | 120 | 122 | 144 | 386
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN | 6 | 10 | 10 | 26
  BLACK OR AFRICAN AMERICAN | 6 | 3 | 4 | 13
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 0 | 1 | 0 | 1
  OTHER | 8 | 8 | 6 | 22
  WHITE | 231 | 231 | 233 | 695

OUTCOME MEASURES:

1. Primary Outcome: RSVPreF3 Specific Immunoglobin (Ig)G Antibody Concentrations Expressed as Group Geometric Mean Concentration (GMC)
Description: Enzyme-linked immunosorbent assay (ELISA) was used to assess the concentrations of IgG antibodies against RSV PreF3 in serum samples.
Time Frame: At 30 days post-vaccination (Day 31)
Population: The analysis was performed on the Per Protocol set (PPS) which consisted of all eligible subjects who received the study intervention as per protocol, had immunogenicity results pre- and post dose, complied with blood draw intervals, without intercurrent conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Units/milliliter
Arm/Group | RSV OA_Lot 1 | RSV OA_Lot 2 | RSV OA_Lot 3
Number analyzed (Participants) | 234 | 237 | 237
ELISA Units/milliliter | 86039.9 [78541.5 to 94254.3] | 80518 [73150 to 88628.2] | 94260.9 [86042.2 to 103264.7]
Statistical Analysis 1: Comparison: RSV OA_Lot 1 vs RSV OA_Lot 2; To demonstrate the clinical equivalence of RSV OA_Lot 1 versus RSV OA_Lot 2 in terms of RSV PreF3 IgG concentrations expressed as group GMC ratio at one month post vaccination. The 2-sided 95% CI for group GMC ratio was derived from an ANCOVA model on log10 transformed RSV PreF3 IgG antibody titers. The ANCOVA model included the treatment group and the age category (age at vaccination: 60-69, 70-79 or >=80 years) and the center as fixed effects and the pre-dose log10 titer as covariate; Test type: Equivalence — Clinical equivalence is demonstrated if the 2 sided 95% confidence interval (CI) of the GMC ratios (RSV OA_Lot 1 divided by RSV OA_Lot 2) is within the pre defined limit of [0.67, 1.5]; Adjusted group GMC ratio = 1.06, 95% CI 2-sided [0.94 to 1.21]
Statistical Analysis 2: Comparison: RSV OA_Lot 1 vs RSV OA_Lot 3; To demonstrate the clinical equivalence of RSV OA_Lot 1 versus RSV OA_Lot 3 in terms of RSV PreF3 IgG concentrations expressed as group GMC ratio at one month post vaccination. The 2-sided 95% CI for group GMC ratio was derived from an ANCOVA model on log10 transformed RSV PreF3 IgG antibody titers. The ANCOVA model included the treatment group and the age category (age at vaccination: 60-69, 70-79 or >=80 years) and the center as fixed effects and the pre-dose log10 titer as covariate; Test type: Equivalence — Clinical equivalence is demonstrated if the 2 sided 95% CI of the GMC ratios (RSV OA_Lot 1 divided by RSV OA_Lot 3) is within the pre defined limit of [0.67, 1.5]; Adjusted group GMC ratio = 0.92, 95% CI 2-sided [0.81 to 1.04]
Statistical Analysis 3: Comparison: RSV OA_Lot 2 vs RSV OA_Lot 3; To demonstrate the clinical equivalence of RSV OA_Lot 2 versus RSV OA_Lot 3 in terms of RSV PreF3 IgG concentrations expressed as group GMC ratio at one month post vaccination. The 2-sided 95% CI for group GMC ratio was derived from an ANCOVA model on log10 transformed RSV PreF3 IgG antibody titers. The ANCOVA model included the treatment group and the age category (age at vaccination: 60-69, 70-79 or >=80 years) and the center as fixed effects and the pre-dose log10 titer as covariate; Test type: Equivalence — Clinical equivalence is demonstrated if the 2 sided 95% CI of the GMC ratios (RSV OA_Lot 2 divided by RSV OA_Lot 3) is within the pre defined limit of [0.67, 1.5]; Adjusted group GMC ratio = 0.87, 95% CI 2-sided [0.77 to 0.99]

2. Secondary Outcome: RSVPreF3 Specific IgG Antibody Concentrations Expressed as Mean Geometric Increase (MGI)
Description: MGI was defined as the geometric mean of the within participant ratios of the post-vaccination RSV PreF3 IgG concentration over the pre-vaccination RSV PreF3 IgG concentration.
Time Frame: At 30 days post-vaccination (Day 31)
Population: The analysis was performed on the PPS which consisted of all eligible subjects who received the study intervention as per protocol, had immunogenicity results pre- and post dose, complied with blood draw intervals, without intercurrent conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | RSV OA_Lot 1 | RSV OA_Lot 2 | RSV OA_Lot 3
Number analyzed (Participants) | 234 | 237 | 237
Ratio | 11.84 [10.53 to 13.31] | 11.29 [10.12 to 12.6] | 12.46 [11.13 to 13.94]

3. Secondary Outcome: Percentage of Participants Reporting Solicited Administration Site Events
Description: Solicited administration site adverse events (AEs) assessed were erythema, pain and swelling. Any = occurrence of the adverse event regardless of intensity grade.
Time Frame: Within 4 days (the day of vaccination and 3 subsequent days) after study intervention administration
Population: The analysis was performed on participants of the Exposed Set (ES) who had their diary cards completed. The ES included all subjects who received the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV OA_Lot 1 | RSV OA_Lot 2 | RSV OA_Lot 3
Number analyzed (Participants) | 249 | 251 | 252
Percentage of participants
  Erythema | 12.4 [8.6 to 17.2] | 11.6 [7.9 to 16.2] | 13.5 [9.5 to 18.3]
  Pain | 58.2 [51.8 to 64.4] | 65.7 [59.5 to 71.6] | 62.7 [56.4 to 68.7]
  Swelling | 6.8 [4 to 10.7] | 7.6 [4.6 to 11.6] | 7.9 [4.9 to 12]

4. Secondary Outcome: Percentage of Participants Reporting Solicited Systemic Events
Description: Solicited systemic events assessed were arthralgia, fatigue, fever [defined as temperature equal to or above (>=) 38 degrees Celsius (°C)/100.4 degrees Fahrenheit (°F)}, headache and myalgia. Any = occurrence of the adverse event regardless of intensity grade or relation to study vaccination.
Time Frame: Within 4 days (the day of vaccination and 3 subsequent days) after study intervention administration
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV OA_Lot 1 | RSV OA_Lot 2 | RSV OA_Lot 3
Number analyzed (Participants) | 249 | 251 | 252
Percentage of participants
  Arthralgia | 13.3 [9.3 to 18.1] | 13.9 [9.9 to 18.9] | 14.7 [10.6 to 19.7]
  Fatigue | 28.1 [22.6 to 34.1] | 25.9 [20.6 to 31.8] | 27.8 [22.3 to 33.7]
  Fever | 2 [0.7 to 4.6] | 1.6 [0.4 to 4] | 2.8 [1.1 to 5.6]
  Headache | 25.7 [20.4 to 31.6] | 23.5 [18.4 to 29.2] | 22.2 [17.2 to 27.9]
  Myalgia | 31.3 [25.6 to 37.5] | 34.3 [28.4 to 40.5] | 33.7 [27.9 to 39.9]

5. Secondary Outcome: Percentage of Participants Reporting at Least One Unsolicited Adverse Event
Description: An unsolicited AE is any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited AE. Unsolicited AEs include serious, non-serious AEs and potential immune-mediated diseases (pIMDs).
Time Frame: Within 30 days (the day of vaccination and 29 subsequent days) after study intervention administration
Population: The analysis was performed on the ES, which included all subjects who received the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV OA_Lot 1 | RSV OA_Lot 2 | RSV OA_Lot 3
Number analyzed (Participants) | 251 | 253 | 253
Percentage of participants | 14.7 [10.6 to 19.7] | 14.6 [10.5 to 19.6] | 13.4 [9.5 to 18.3]

6. Secondary Outcome: Percentage of Participants Reporting at Least One Serious Adverse Event (SAE)
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant. Any = occurrence of the symptom regardless of intensity grade or relationship to vaccination.
Time Frame: From Day 1 up to study end (6 months after vaccination)
Population: The analysis was performed on the ES, which included all subjects who received the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | RSV OA_Lot 1 | RSV OA_Lot 2 | RSV OA_Lot 3
Number analyzed (Participants) | 251 | 253 | 253
Percentage of Participants | 3.2 [1.4 to 6.2] | 2.4 [0.9 to 5.1] | 2.8 [1.1 to 5.6]

7. Secondary Outcome: Percentage of Participants Reporting at Least One Potential Immune-mediated Disease (pIMD)
Description: pIMDs are a subset of AEs of special interest that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
Time Frame: From Day 1 up to study end (6 months after vaccination)
Population: The analysis was performed on the ES, which included all subjects who received the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV OA_Lot 1 | RSV OA_Lot 2 | RSV OA_Lot 3
Number analyzed (Participants) | 251 | 253 | 253
Percentage of participants | 0.8 [0.1 to 2.8] | 0.4 [0 to 2.2] | 1.2 [0.2 to 3.4]

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected during the 4-day follow-up period after vaccination. Unsolicited AEs were collected during the 30-day follow-up period after vaccination. SAEs and pIMDs were collected throughout the study period (from Day 1 to Study end (6 months after vaccination)).
Arm/Group | RSV OA_Lot 1 | RSV OA_Lot 2 | RSV OA_Lot 3
All-Cause Mortality (participants affected / at risk) | 0/251 | 2/253 | 2/253
Serious Adverse Events (participants affected / at risk) | 8/251 | 6/253 | 7/253
Other Adverse Events (participants affected / at risk) | 181/251 | 192/253 | 195/253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV OA_Lot 1 (N=251) | RSV OA_Lot 2 (N=253) | RSV OA_Lot 3 (N=253)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of the hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Large intestine infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV OA_Lot 1 (N=251) | RSV OA_Lot 2 (N=253) | RSV OA_Lot 3 (N=253)
Injection site pain (General disorders) | 145 (145) | 165 (165) | 159 (160)
Fatigue (General disorders) | 70 (70) | 66 (66) | 72 (72)
Injection site erythema (General disorders) | 32 (32) | 29 (29) | 37 (37)
Injection site swelling (General disorders) | 17 (17) | 20 (20) | 20 (20)
Pyrexia (General disorders) | 8 (8) | 9 (9) | 9 (9)
Chest discomfort (General disorders) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Tenderness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 78 (78) | 87 (87) | 86 (86)
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 (34) | 36 (37) | 39 (39)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 65 (68) | 62 (64) | 57 (59)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Ophthalmic migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis caliciviral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral mucosal blistering (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Age-related macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Computerised tomogram head abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT05059301/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT05059301/SAP_001.pdf